CLINICAL TRIAL: NCT05464316
Title: Comparing the Effectiveness of the Adjustable Trans Obutator Male System (ATOMS) Versus the Artificial Urinary Sphincter (AUS) in Moderate to Severe Post-Prostatectomy Stress Urinary Incontinence
Brief Title: Prospective Pilot ATOMS vs AUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Le Mai Tu, Urologist, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-4477
Record Dates: First submitted 2022-06-28; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Post-Prostatectomy Incontinence; Urinary Stress Incontinence; Urinary Incontinence; Stress Incontinence, Male
Keywords: ATOMS; AUS; Prospective
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence | interventions — Urinary Sphincter, Artificial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjustable Transobturator Male System (Experimental)
  Interventions: Device: Adjustable Transobturator Male System
- Artificial Urinary Sphincter (Active Comparator)
  Interventions: Device: Artificial Urinary Sphincter

INTERVENTIONS:
Device: Adjustable Transobturator Male System — The ATOMS sling was developed in 2008 by Agency for Medical Innovations GmbH in Austria. It is a self-anchoring adjustable system which supports the bulbar urethra dorsally and uses the trans obturator approach. This device gained its fame in the male sling scene by being adjustable, which theoretically makes it more efficacious than its competitors.
  Arms: Adjustable Transobturator Male System
Device: Artificial Urinary Sphincter — The AMS800™, which is by far the most frequently implanted AUS, was first marketed in 1983 and was developed by America Medical Holdings in Minnesota. Today, the AUS has been given the title "gold standard" for surgical treatment for PPI. This device is an inflatable cuff which wraps around the urethra to supply circumferential pressure. It has a control pump, which is found in the scrotum and is operated by the patient. The patient can void simply by squeezing the pump, which brings the fluid from the cuff to a reservoir and release the pressure around the urethra. The cuff is then automatically refilled with fluid within a couple of minutes to close back the sphincter.
  Arms: Artificial Urinary Sphincter

SUMMARY:
Post-Prostatectomy Incontinence (PPI) is a common complication affecting 1% to 40% of patients after surgery. When conservative treatments fail, the installation of an artificial urinary sphincter (AUS) has been the treatment of choice for PPI since its introduction more than 50 years ago. Although small studies suggest inferior success rate of male slings compare to the AUS in moderate to severe male incontinence; recent studies, one prospective and one Canadian multicenter cohort study, have demonstrated adjustable transobturator male sling (ATOMS) as a safe and efficient alternative to treat PPI. Interestingly, the ATOMS does not required any operation manipulation from the user in order to void and it causes potentially less urethral erosion and less urethral atrophy than the AUS; although those findings were never compared head to head with the AUS. Therefore, we believe that a thorough prospective non-inferiority study comparing the outcomes and effectiveness of the ATOMS device versus the AUS in treating moderate to severe PPI could prove itself useful in guiding urologists and patients to choose their best treatment of male incontinence. The null hypothesis posed for the present study is that ATOMS is non inferior to AUS for the treatment of moderate to severe PPI using the non-inferiority margin of 15% to be of acceptable lower effectiveness.

With regards to study methods, this will be a pilot prospective, randomized controlled trial, non-blinded with a non-inferiority design. This pilot study will take place at the CIUSSS de l'Estrie, in Sherbrooke, Quebec, Canada, with two surgeons. All male patients with moderate to severe incontinence after their prostate surgery, who are suitable for incontinence surgery will be screened for study eligibility respecting the exclusion and inclusion criteria. After written informed consent, enrolled patients will be randomized assigned (1:1) to one of the two interventions' arms (AUS or ATOMS). Sixty patients are estimated to be randomized in the two arms the day of their surgery with a computer-based algorithm sequence.

By completing this pilot prospective study, we hope to provide concrete and scientifically significant evidence on the effectiveness of ATOMS in the treatment of moderate to severe PPI comparing with the AUS. Although both treatments are commonly used today, there has been little evidence comparing both devices side by side with more severe PPI. We therefore hope to make a global impact with said project.

ELIGIBILITY:
Inclusion Criteria:

* Adult men (≥ 18 years of age) with moderate-to-severe post-prostatectomy urinary incontinence who are eligible and have consented to receive surgery as treatment. Determining patient eligibility for surgery is based on the AUA/SUFU Guidelines, published in 2019.
* Patients who consented to being randomised in receiving ATOMS and AUS.

Exclusion Criteria:

* Patients whom the physician determines to be poor candidates for surgical procedures and/or anesthesia due to; poor manual dexterity, poor cognitive function, and other physical or mental conditions.
* Patients who have unresolved urethral or urethral-vesical anastomose stenosis within the last 12 months.
* Patients who have undergone previous incontinence surgeries.
* Patients who suffer mild incontinence (less than 200g per day).
* Patients with primarily neurogenic incontinence.
* Patients with rising PSA levels within the previous 12 months.
* Patients with urinary incontinence due to or complicated by an irreversibly obstructed lower urinary tract"
* Patients with known allergies or sensitivity to rifampin or to minocycline HCl or other tetracyclines.", in InhibiZone implantation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-01-13 (Estimated); Study Completion 2025-01-13 (Estimated)

PRIMARY OUTCOMES:
To compare effectiveness of the ATOMS and AUS devices in patients using results from the Patient Global Impression of Improvement (PGI-I) questionnaire. | Three years
To compare effectiveness of the ATOMS and AUS devices in patients using results from the 24-hour pad test. | Three years

SECONDARY OUTCOMES:
To compare complication rates of the AUS and ATOMS using the Clavien-Dindo Classification. | Three years
To compare effectiveness of the AUS and ATOMS devices in patients using results from the ICIQ-UI SF questionnaire. | Three years
To compare effectiveness of the AUS and ATOMS devices in patients using results from the ICIQ-OAB questionnaire. | Three years
To compare effectiveness of the AUS and ATOMS devices in patients using results from the ICIQ-MLUTS LF questionnaire. | Three years
To compare effectiveness of the AUS and ATOMS devices in patients using results from the IPSS-QoL questionnaire. | Three years
To assess the impact of OAB and radiotherapy on the effectiveness of AUS and ATOMS using results from the Patient Global Impression of Improvement (PGI-I) questionnaire. | Three years
To assess the impact of OAB and radiotherapy on the effectiveness of AUS and ATOMS using results from the 24-hour pad test. | Three years
To assess the impact of OAB and radiotherapy on the safety of AUS and ATOMS using Clavien-Dindo Classification to report adverse event frequency and severity. | Three years
To assess the impact of OAB and radiotherapy on the effectiveness of AUS and ATOMS using results from the ICIQ-UI SF questionnaire. | Three years
To assess the impact of OAB and radiotherapy on the effectiveness of AUS and ATOMS using results from the ICIQ-OAB questionnaire. | Three years
To assess the impact of OAB and radiotherapy on the effectiveness of AUS and ATOMS using results from the ICIQ-MLUTS LF questionnaire. | Three years
To assess the impact of OAB and radiotherapy on the effectiveness of AUS and ATOMS using results from the IPSS-QoL questionnaire. | Three years
To assess the impact of OAB and radiotherapy on the effectiveness of AUS and ATOMS using results from the 24-hour pad-count. | Three years
To compare effectiveness rates of the AUS and ATOMS using the results of the 24-hour pad-counts. | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fleurimont- Centre Hospitalier de l'Université de Sherbrooke, Sherbrooke, Quebec, Canada